CLINICAL TRIAL: NCT05833945
Title: Study of the Potential Use of a Rapid Point-of-Care Device for the Direct Transfer of Stroke Patients From the Ambulance to the Thrombectomy Center
Brief Title: Potential Use of a POCT for the Direct Transfer of Stroke Patients From the Ambulance to the Thrombectomy Center
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Hospital Universitario Virgen Macarena (Other); Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Torrecárdenas (Other); Hospital Universitario Poniente (Unknown); Hospital Clínico Universitario Lozano Blesa (Other); Hospital Miguel Servet (Other); Hospital Universitario Royo Villanova (Unknown); Hospital General San Jorge (Unknown); Hospital San Pedro de Logroño (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Universitario La Fe (Other); Complejo Hospitalario Universitario de Albacete (Other); Hospital de Medina del Campo (Unknown); Hospital General Río Carrión (Unknown); Hospital General de Segovia (Other); Hospital del Rio Hortega (Other)
Responsible Party: Sponsor
Other Study IDs: BIOSHIP-training
Record Dates: First submitted 2023-04-05; First posted 2023-04-27 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Stroke, Acute Ischemic
Keywords: Large Vessels Occlusion (LVO); Thrombectomy; Biomarkers; Point of care test (POCT)
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-hospital and in-hospital patients: Patients recruited at the ambulance (ARM A) and at the hospital (ARM B).
  Interventions: Device: Large Vessel Occlusion Biomarkers Test

INTERVENTIONS:
Device: Large Vessel Occlusion Biomarkers Test — Duplex Point of Care test to measure the concentration of biomarkers associated to Large Vessel Occlusion in blood samples used in combination with an APP.

SUMMARY:
Stroke is the leading cause of long-term disability and the second most common cause of death worldwide. Currently, the protocols require the imaging techniques at the hospitals to differ ischemic strokes with large vessel occlusion (LVO) from others. In this study, a duplex POC will be used in combination with an APP to identify LVO ischemic strokes in a 800 patients'cohort with pre-hospital and in-hospital blood samples.

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability and the second most common cause of death worldwide, accounting for around 6.7 million deaths each year. The burden of stroke due to illness, disability and early death is set to double within the next 15 years due to an ageing population. Currently, imaging techniques are required to differentiate ischemic strokes with large vessel occlusion (LVO) from others. Since those neuroimages cannot be easily done at a pre-hospital level, our objective is to develop a simple point-of-care test (POC) to differentiate between both ischemic strokes during the acute phase, which will allow in the future an earlier thrombectomy treatment and an improvement of the patient outcomes significantly. For that, the investigators will recruit a 800 patients' cohort with pre-hospital and in-hospital blood samples by a multiplex POC for the biomarker measurement using an APP in combination with clinical data to identify LVO ischemic strokes. Finally, an interim analysis is planned when 400 patients are recruited.

ELIGIBILITY:
Inclusion Criteria:

* I.1: Patients > 18 years old.
* I.2: Stroke code activated.
* I.3: < 6 hours from symptoms onset. In the case of stroke with uncertain chronology or wake-up stroke, the initial time will be considered as the last moment the patient was seen fine.

Exclusion Criteria:

* E.1: Previous diagnosis different from stroke.
* E.2: Impossibility of getting a blood sample.
* E.3: Refusal to provide the informed consent by the patient/relative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke code activated will be recruited at a pre-hospital and hospital environment.
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diagnosis accuracy of the algorithm LVOCheck (Specificity and sensibility) | 6 months
  * Biomarkers
  * Clinical data (gender, age, diabetes, dyslipidemia, atrial fibrillation, blood pressure)
  * Neurologic scales (NIHSS, RACE, GFAST, Cincinatti)

SECONDARY OUTCOMES:
Viability of the implement of the tool at a pre-hospital environment | 6 months
  * Estimated time in patients direct potentially transferred to the thrombectomy centers.
  * Error rate in tool performance at a pre-hospital and hospital environment.
  * Percentage of right use of the tool (human failares) at a pre-hospital and hospital environment.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Barragán Prieto, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (16):
- Spain (16):
  - Complejo Hospitalario Universitario Albacete, Albacete
  - Hospital Universitario Poniente, Almería
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital General San Jorge, Huesca
  - Hospital San Pedro, Logroño
  - Hospital General Río Carrión, Palencia
  - Hospital General de Segovia, Segovia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Rocío, Seville
  - Hospital La Fe, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital de Medina del Campo, Valladolid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza
  - Hospital Royo Villanova, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) might be included in a publication. Specific data set are not determined yet.